CLINICAL TRIAL: NCT06147102
Title: The Helsinki Unruptured Intracranial Aneurysm Quality of Care Study
Acronym: HUIQE
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Rahul Raj, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: HUS/216/2023
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysm; surgery; neurosurgery; endovascular; interventional neuroradiology; neurointervention; unruptured
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular treatment: Patients with unruptured intracranial aneurysms treated endovascularly
  Interventions: Procedure: Endovascular
- Surgical treatment: Patients with unruptured intracranial aneurysms treated surgically
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgical treatment for the unruptured intracranial aneurysm
  Groups: Surgical treatment
Procedure: Endovascular — Endovascular treatment for the unruptured intracranial aneurysm
  Groups: Endovascular treatment

SUMMARY:
A research-initiated prospective cohort study with the aim to assess the effectivity, safety and long-term outcomes after surgical and endovascular treatment of unruptured intracranial aneurysms. All consecutive patients with a non-ruptured intracranial aneurysms treated at Helsinki University Hospital will be included. Safety is measured by postoperative magnetic resonance imaging (MRI) taken 1-3 days after the treatment, treatment-related complications and functional outcome at three months. Effectiveness is measured by angiographic results and assessment of long-term bleeding from the treated aneurysm. Other outcomes include risk of developing epilepsy, getting a new stroke, and dementia on long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an unruptured intracranial aneurysm undergoing treatment

Exclusion Criteria:

* Arteriovenous malformation related intracranial aneurysm
* Moyamoya-disease related intracranial aneurysm
* Ruptured intracranial aneurysm

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing endovascular or surgical treatment for an unruptured intracranial aneurysm at Helsinki university hospital
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
New ischemic lesion on postoperative MRI | 1-3 days
  Diffusion-Weighted Imaging lesion

SECONDARY OUTCOMES:
Neurological symptom | 3 months
  New procedure-related neurological symptom
Return to work | 3 months
  Days from intervention to return to work
Functional outcome | 3 months
  modified Rankin Scale (mRS going from 0 [no sympyoms] to 6 death])
Aneurysm occlusion on angiography | 6mo - 5yrs
  Rate of occluded vs. incompletely occluded aneurysms. Assessed through digital subtraction angiography, CTA or MRA. Routine controls for endovascularly treated patients 6mo, 2y, and if needed 5y. Routinely assessed by a postoperative CTA for surgically treated patients.
Patients with late rebleeding from the target aneurysm | up to 10 yrs
  Number of patients with rebleeding (subarachnoid hemorrhage [SAH]) from the treated aneurysm
Epilepsy | up to 10 yrs
  Number of patients with a new diagnosis of epilepsy after aneurysm treatment
Dementia | up to 10 yrs
  Number of patients with a new diagnosis of dementia after aneurysm treatment
Other stroke than aneurysm bleed | up to 10 yrs
  Number of patients with a new stroke (other than SAH from the treated aneurysm) after aneurysm treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Raj, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing regulated by the Secondary Use of Health And Social Data Act in Finland.

REFERENCES:
- [Derived] Raj R, Numminen J, Huhtakangas J, Nurminen V, Lehecka M, Laakso A, Kivipelto L, Niemela M, Korja M. The Helsinki Unruptured Intracranial Aneurysm Quality of Care study: a prospective observational study. J Neurosurg. 2025 Dec 5:1-10. doi: 10.3171/2025.7.JNS25775. Online ahead of print. PMID 41349033